CLINICAL TRIAL: NCT03100513
Title: Randomized Trial Comparing The Efficacy of PEG (Polyethylene Glycol) Versus Lactulose For Treatment Of Overt Hepatic Encephalopathy
Brief Title: PEG (Polyethylene Glycol)Versus Lactulose For Treatment Of Overt Hepatic Encephalopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Clinical Ass Prof. Hepatology and Gastroenterology, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hanan Soliman
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactulose (Active Comparator): (20 to 30 g administered orally or by nasogastric tube (3 or more doses within 24 hours) or 200 g by rectal tube if oral intake was not possible or inadequate.
  Interventions: Drug: Lactulose
- Polyeyhylene Glychol (Active Comparator): Polyethylene Glycol 3sachets if patient <75Kg over 3 hours or 4 sachets if patient >75Kg over 4 hours dministered orally or via a nasogastric tube (each sachet 64g/25Kg must be dissolved in one liter of water)
  Interventions: Drug: Polyethylene Glycol

INTERVENTIONS:
Drug: Lactulose — (lactulose) (20 to 30 g administered orally or by nasogastric tube (3 or more doses within 24 hours) or 200 g by rectal tube if oral intake was not possible or inadequate
  Other Names: Duphlac, lactulose
  Arms: Lactulose
Drug: Polyethylene Glycol — PEG as single dose of (3sachets if patient <75Kg over 3 hours or 4 sachets if patient >75Kg over 4 hours) dministered orally or via a nasogastric tube (each sachet 64g/25Kg must be dissolved in one liter of water).
  Arms: Polyeyhylene Glychol

SUMMARY:
The current standard of care for patients with HE includes non-absorbable disaccharides(lactulose);The chemical name for lactulose is 4-O-β-D-galactopyranosyl-D-fructofuranose.The exact mode of action by lactulose is thought to be the conversion to lactic acid and acetic acid by colonic bacteria resulting in acidification of the gut lumen. This favors conversion of ammonia (NH3) to ammonium (NH4+), which is relatively membrane impermeable; therefore, less ammonia is absorbed by the colon. Gut acidification inhibits ammoniagenic coliform bacteria, leading to increased levels of nonammoniagenic lactobacilli. Nonabsorbable disaccharides also work as a cathartic, clearing the gut of ammonia before it can be absorbed.

DETAILED DESCRIPTION:
Polyethylene glycol electrolyte solution (PEG) is a laxative solution that increases the amount of water in the intestinal tract to stimulate bowel movements. It is used safely to clean the bowel before colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with Overt Hepatic Encephalopathy.

Exclusion Criteria:

1. Patients with active GIT bleeding.
2. Patients with history of bowel obstruction, perforation.
3. Patients with history of allergy to PEG.
4. Treatment with rifaximin or neomycin in the previous 7 days.
5. Patients with major psychiatric illness.
6. Patients receiving benzodiazepines and narcotics.
7. Patients with compromised renal.
8. Patients receiving medications highly bound to plasma proteins eg. Warfarin.
9. Pregnant or lactating women.
10. Fulminant hepatic failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-11 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
1 or more in HE grade improvement at 24 hours | 24 hours
  HE grade improvement at 24 hours

SECONDARY OUTCOMES:
Time to HE resolution | 2 weeks
  Time to Hepatic encephalopathy resolution
Overall length of stay | 2 weeks
  Overall length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Soliman, MD, Principal Investigator — Tanta University Faculty of Medicine; Amany Abd El-Rahim Abdin, MD, Study Director — Tanta university Faculty of Pharmacy; Samah Mosaad Soliman, MD, Study Director — Tanta University Faculty of Medicine; Hala Hany Shehata, Msc, Study Chair — Tanta University Faculty of Medicine; Sherief Abd-Elsalam, MD, Study Chair — Tanta University Faculty of Medicine
Locations (1):
- Tropical medicine dept.-Tanta university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided